CLINICAL TRIAL: NCT04300868
Title: Immunisation Status Against Major Communicable Diseases Preventable With Vaccines, and Safety of Vaccines, in a Cohort of MS Patients. An Italian Multicenter Study
Brief Title: Immunisation Status and Safety of Vaccines in Italian MS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Monica Ulivelli (Other)
Collaborators: Fondazione Italiana Sclerosi Multipla (Other); San Luigi Gonzaga Hospital (Other); University of Roma La Sapienza (Other); Universita degli Studi di Catania (Other); Universita degli Studi di Genova (Other); San Camillo Hospital, Rome (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); University of Florence (Other); Istituto Neurologico Mediterraneo Neuromed S. R. L (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Maggiore Bellaria Hospital, Bologna (Other); Federico II University (Other); Ospedale San Donato (Other); Ospedale San Giuseppe di Empoli (Other); Ospedale Livorno (Other); Ospedale Misericordia e Dolce (Other); Ospedale della Misericordia (Other); Ospedale San Jacopo (Unknown); Ospedale Felice Lotti di Pontedera (Other); Campus Bio-Medico University (Other); Università degli Studi di Ferrara (Other)
Responsible Party: Sponsor-Investigator, Monica Ulivelli, researcher, University of Siena
Organization: University of Siena (Other)
Other Study IDs: 2019/S/2
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
Keywords: immunisation status; vaccine safety; vaccination
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple sclerosis (MS) patients are more susceptible to infections than the general population in relation to some specific therapies or increasing disability. Clearly, the use of immuno-suppressant/modulatory drugs requires particular attention to the occurrence of infectious events. In this perspective, among still unmet clinical needs in MS patients is a comprehensive picture on the immunisation status against infectious diseases, especially those preventable with vaccines. Despite of the relevance of vaccinations, there are still some concerns about their utilization in MS patients. In literature, results about their safety are conflicting or incomplete and it is yet unclear if some vaccines may trigger MS relapses.

GOALS: 1) to assess immunisation status, due to past exposure to natural infectious diseases or vaccines, against major infectious agents preventable by available vaccines; 2) to assess the safety of most utilized vaccines in the clinical practice by recording relapses as adverse event in the considered risk period after vaccination.

The 3-year project is conceived as a multicenter, observational, both retro- and prospective study. A cohort of about 3,000 MS subjects will be enrolled among databases of 25 clinical Centers in Italy. All patients diagnosed with relapsing remitting (RR) MS according to the 2010 Polman's criteria from 01/2011 to 12/2020 will be enrolled. Available data on natural immunisation will be collected from the historical clinical records of Centers, taking into account the presence of specific serum antibodies, whereas available data on vaccinations will be collected from vaccination records.

To study the impact of vaccines on the risk of relapse, data about patients receiving a vaccination during the disease will be analysed. The study follow-up period will be between 2 and up to 6 months following vaccination: the 2-month period is considered as the maximum clinical risk, whereas 6 months as the maximal extension of risk in time. In addition, in the case of a clinical relapse, the variation of disability will be evaluated with EDSS scale confirmed at 6 months. These data might shed light on the relationship between vaccination and MS, adding new insights on their safety.

The knowledge of the immunisation status is crucial for the clinical practice in the management of the new disease modifying drugs (DMDs), and for the public health to establish the possible need of a vaccine campaign targeted to MS patients.

DETAILED DESCRIPTION:
The different available treatments for MS influence the immune system in distinct ways and, therefore, may lead to specific infectious risks. Whereas immunomodulating therapies have no impact on infection risks [Cahill 2010; Winkelmann 2016], the most recent drugs with immunosuppressant activity could increase persons with MS' vulnerability to infections [Löbermann 2012; Olsson 2014]. MS patients are routinely screened for latent or active infections before starting any disease modifying drugs (DMDs). Specific infectious agents should be evaluated for each second line [Williamson 2015, Yang 2014, Kohlmann 2015]. Another cause of increased susceptibility to infections in MS patients is disability: patients have a greater risk for serious and fatal infections due to MS-related functional limitations as pulmonary problems and bladder and bowel dysfunctions [Montgomery 2013; Nelson 2015]. In addition, there is consistent evidence that exacerbations could be a consequence of infectious diseases, such as bacterial infections of urinary tract, viral respiratory diseases or gastroenteritis, with a two-fold increase in risk of relapse after infection [Panitch 1994; Rutschmann 2002; Loebermann 2012; Williamson 2015]. In such case, the mechanisms underlying relapses are not fully understood [Steelman 2015], but probably molecular mimicry and bystander activation play a role in this process [Loebermann 2012]. Therefore, it is important to promote any prevention strategy that may reduce the risk of acquiring infections, such as vaccination.

Vaccination is the main proven tool for primary prevention of serious, and sometimes life-threatening diseases and one of the most cost-effective public health measures available.

There are 4 main types of vaccines: live-attenuated vaccines, inactivated vaccines, subunit/recombinant/polysaccharide/conjugate vaccines and toxoid vaccines. Live vaccines are made using an attenuated or weakened form of the pathogen. These vaccines have a high efficacy but, containing a live pathogen, they have a potential risk of infection, particularly in patients with a natural or acquired immunodeficiency. Further, concerns about live vaccines administration to close family members of patients have been raised, as there could be the risk that immunised individual release the live pathogens [Williamson 2016]. On the contrary, the other types of vaccines can be safely used by persons with an impaired immune system [www.vaccines.gov].

In Italy, before 2017, 4 vaccinations were mandatory for children (against diphtheria from 1939, polio from 1966, tetanus from 1968 and hepatitis B from 1991), whereas several others were only recommended. Due to inadequate immunisation coverage, the obligation was recently extended to 10 vaccines, adding the ones against Haemophilus influenzae type B, pertussis, measles, mumps, rubella and varicella for newborns. In addition, there are other recommended vaccines at different ages, i.e. vaccination against rotavirus, meningitis B and C, pneumococcal disease in childhood, against human papilloma virus in adolescents, and against tetanus, diphtheria, pertussis, influenza, pneumococcal disease and herpes zoster for those aged 65 years and older [www.salute.gov.it].

In MS population, there are some concerns about the utilization of vaccines. It is unclear (at least for some vaccines) whether vaccinations may trigger the disease or increase the risk of relapse due to the stimulation of the immune system, as the infections themselves [Loebermann 2012]. The vaccines against hepatitis B virus, tetanus, tick-borne encephalitis, H1N1 virus and seasonal influenza are considered safe, even if small groups of patients (with a very active form of MS) report an increased risk of relapse after influenza or H1N1 vaccine [Loebermann 2012]. An increased risk of relapses was reported also after yellow-fever immunisation in a single study conducted in a very small cohort of RR-MS patients [Farez 2011b]. On the other hand, a protective role is reported for some vaccines, for example for bacillus Calmette-Guérin vaccine, and for vaccines against tetanus and diphtheria [Loebermann 2012]. For all other vaccines, no data are available [Mailand 2017].

Moreover, specific DMDs may increase the risk of infectious complications from vaccines composed by live attenuated microorganism [MSC for clinical practice guidelines]. Live attenuated vaccines are considered safe for patients receiving an immunomodulator agent such as glatiramer acetate or interferon, but there are relatively few data on the safety of these vaccines for the more recently approved immunosuppressant agents. Hence, patients treated with these drugs should avoid live attenuated vaccines during the treatment and for a period of 3 months after discontinuation of treatment [Cahill 2010; Oreja-Guevara 2014]. In addition, MS patients experiencing a serious relapse should delay the vaccination until 4-6 weeks after the exacerbation [National MS society].

Finally, DMDs could reduce the efficacy of vaccination leaving people susceptible to diseases, however the published studies showed conflicting results [Williamson 2016].

Several new drugs have been developed to treat multiple sclerosis (MS) in the last 2 decades. Balancing benefit and risk in recent MS treatment management is decisive. In the era of disease modifying drugs (DMDs), that alter immune function, the reactivation or de novo acquisition of infectious diseases is gaining great relevance. The understanding of the potential adverse effects of these immunological active therapies is a key part of the decision-making process when weighting different treatment options. Consequently, prior to starting an immunosuppressant treatment, it is necessary to know the immunisation status of patients, including immunity elicited both by natural infections and vaccinations. The knowledge of susceptibility to infections of patients is recommended for therapeutic choice.

First of all, it is mandatory for some immunosuppressant drugs, or suggested for others, to assess the immunisation status against herpes zoster virus, because the reactivation of this disease might be serious. Vaccinations against varicella and herpes zoster contain the live-attenuated virus, so immunocompromised patients should not be immunised with these vaccines [Williamson 2016]. For the same reason, the immunisation against measles, mumps and rubella could be recommended in susceptible subjects because these pathogens could trigger serious complications, such as encephalitis and pneumonia. Therefore, in patients who have never had natural infections, it could be necessary to take into account immunisation with these live-attenuated vaccines just early after MS diagnosis, in view of a possible future treatment with an immunosuppressant drug.

In addition, there are other vaccines against other frequent infectious agents which are recommended for general population and for groups at risk: tetanus, diphtheria and pertussis (which require a booster dose every 10 years for all persons), seasonal influenza, pneumococcal, meningococcal, Haemophilus influenzae type B (Hib), hepatitis A and B virus. According to the international public health recommendations, all individuals in the older age groups (usually over 65 years of age) and those from age of 6 months with a chronic disease with increased risk for severe outcomes of influenza complications, must be vaccinated every year. The medical conditions that could represent a risk factor for influenza complications include any situation compromising respiratory functions, as in many neurological disorders, and the immunosuppression due to disease or treatment [www.ecdc.europa.eu]. For the same reasons, the pneumococcal vaccine is recommended because, in susceptible people, flu virus may trigger an infection by Streptococcus pneumoniae [www.cdc.gov]. Regarding Hib, individuals with a secondary immunodeficiency may be at risk of developing invasive disease if exposed to the pathogen [Nix 2012]. In case of outbreak of meningococcal or hepatitis A, or in case of risk of hepatitis B, adults might be vaccinated [www.ecdc.europa.eu].

Another aspect to take into account is the presence of hepatitis B chronic infections, as the immunosuppressant treatment must be preceded and accompanied by a specific antiretroviral drug blocking the viral DNA synthesis [Orlicka 2013].

The positive effect on individual well being is coupled with a favourable economic impact in public health. Also in patients with MS, vaccination could reduce the disease burden and consequently the social cost, as it might reduce eventual relapses or other severe complications [Rutschmann 2002]. Therefore, the knowledge of the immunisation status could help policy makers and program strategies to assess the need of a vaccine campaign targeted to MS patients.

Despite these considerations, there are no available data about the prevalence of patients susceptible to infections, therefore unvaccinated or people never exposed to natural infections. Concerning the severe and potentially life-threatening infective complications associated with the immunosuppressant agents used to treat MS, the use of specific registries and databases to collect and evaluate infection/vaccine safety data after drug approval is advisable.

The safety of most vaccines in MS patients has been only partly investigated, so that a correlation between vaccination and MS relapses has been hypothesized only for some vaccines. However, these conclusions are based on few studies, mostly carried out on small study sample sizes. The lack of large amounts of data regarding the vaccine safety in MS population precludes the possibility to offer clear-cut recommendations.

The first aim of the study is to collect historical data on the immunisation status, due to past exposure to natural infectious diseases or vaccines, in a large multicentric cohort of MS patients with regards to the most frequent vaccine-preventable viral and bacterial infections.

The second aim is to assess the potential role of vaccines used in adulthood in determining/worsening MS inflammatory activity, as well in disease progression. In particular, any vaccination against hepatitis A and B, measles, mumps, rubella, varicella, diphtheria, pertussis, seasonal influenza, herpes zoster virus, meningococcal and pneumococcal bacteria will be considered. In addition to these communicable diseases, the tetanus vaccine will be included due to the high coverage of this vaccination. MS activity and progression will be assessed evaluating the occurrence of relapse within 6 months from vaccination and using the annual relapse rate and its trend during the study period.

STUDY DESIGN The project is a 3-year observational, retro- and prospective study. Aim 1: Multicenter cross-sectional study on the immunisation status, due to past exposure to natural infectious diseases or vaccines, will be conducted in a MS patient cohort. Sub-analyses will be stratified by sex, patient's age at the time of enrolment, disease duration from clinical onset, disability, current/past DMDs, geographic area of birth and residence, type of vaccine, comorbidity with special regard to autoimmune/immune mediated and/or infectious diseases. 25 MS Centers from Northern, Central and Southern Italy will represent the study sites.

Aim 2: The potential role of vaccines used in adulthood in determining/worsening MS inflammatory activity, as well on disease progression will be conducted by means of a self-controlled case series study over the all MS cohort. A 'case' will be defined as 'exposed' if at least one confirmed relapse occurred during the risk period of 2 months and during the extended risk period of 6 months after vaccine administration; and not exposed otherwise [Galeotti 2013].

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of RR-MS according to the 2010 Polman's diagnostic criteria [Polman 2011] or the 2017 revision of the McDonald criteria for the prospective cohort [Thompson 2018]
* written informed consent must be obtained before the enrolment

Exclusion Criteria:

* clinically isolated syndrome (CIS) and progressive MS forms
* unavailability or unreliability of medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsing remitting (RR)-MS patients consecutively diagnosed from January 2011 to December 2020 will be enrolled in the study upon informed written consent. The choice of January 2011 is suggested by the need to apply the 2010 Polman's diagnostic criteria for MS [Polman 2011] in order to ensure most homogeneous diagnoses across patients.
  Both for retrospective and prospective phase, each Center will identify, through clinical records, newly diagnosed MS patients in the considered period and consistently followed in the Center, and the enrolment will be made during routine ambulatory visits.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of MS patients susceptible to infections | december 2021
  prevalence of patients unvaccinated or never exposed to natural infections, which can represent a problem in case of administration of immunosuppresive drugs.

SECONDARY OUTCOMES:
safety of vaccination in MS patients | december 2021
  evaluation of safety of vaccination in MS patients, considering the occurrence of relapses or a progression of disability 2-6 months after a vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Monica Ulivelli, researcher, Principal Investigator — University of Siena
Locations (1):
- university of Siena, Siena, SI, Italy

REFERENCES:
- [Background] Cahill JFX, Izzo A, Garg N (2010) Immunisation in patients with Multiple Sclerosis. Neurol. Bull, 2:17-21. 10.7191/neurol_bull.2010.1020
- [Background] Farez MF, Correale J. Yellow fever vaccination and increased relapse rate in travelers with multiple sclerosis. Arch Neurol. 2011 Oct;68(10):1267-71. doi: 10.1001/archneurol.2011.131. Epub 2011 Jun 13. PMID 21670384
- [Background] Galeotti F, Massari M, D'Alessandro R, Beghi E, Chio A, Logroscino G, Filippini G, Benedetti MD, Pugliatti M, Santuccio C, Raschetti R; ITANG study group. Risk of Guillain-Barre syndrome after 2010-2011 influenza vaccination. Eur J Epidemiol. 2013 May;28(5):433-44. doi: 10.1007/s10654-013-9797-8. Epub 2013 Mar 31. PMID 23543123
- [Background] Kohlmann R, Salmen A, Chan A, Knabbe C, Diekmann J, Brockmeyer N, Skaletz-Rorowski A, Michalik C, Gold R, Uberla K. Serological evidence of increased susceptibility to varicella-zoster virus reactivation or reinfection in natalizumab-treated patients with multiple sclerosis. Mult Scler. 2015 Dec;21(14):1823-32. doi: 10.1177/1352458515576984. Epub 2015 Mar 31. PMID 25828755
- [Background] Lobermann M, Borso D, Hilgendorf I, Fritzsche C, Zettl UK, Reisinger EC. Immunization in the adult immunocompromised host. Autoimmun Rev. 2012 Jan;11(3):212-8. doi: 10.1016/j.autrev.2011.05.015. Epub 2011 May 18. PMID 21621004
- [Background] Loebermann M, Winkelmann A, Hartung HP, Hengel H, Reisinger EC, Zettl UK. Vaccination against infection in patients with multiple sclerosis. Nat Rev Neurol. 2012 Jan 24;8(3):143-51. doi: 10.1038/nrneurol.2012.8. PMID 22270022
- [Background] Mailand MT, Frederiksen JL. Vaccines and multiple sclerosis: a systematic review. J Neurol. 2017 Jun;264(6):1035-1050. doi: 10.1007/s00415-016-8263-4. Epub 2016 Sep 7. PMID 27604618
- [Background] Montgomery S, Hillert J, Bahmanyar S. Hospital admission due to infections in multiple sclerosis patients. Eur J Neurol. 2013 Aug;20(8):1153-60. doi: 10.1111/ene.12130. Epub 2013 Mar 16. PMID 23496086
- [Background] MS council for clinical practice guideline. Immunisation and multiple sclerosis. Evidence-Based Management Strategies for Immunisations in Multiple Sclerosis. Nov 2001
- [Background] National MS society Vaccinations https://www.nationalmssociety.org/Living-Well-With-MS/Diet-Exercise-Healthy-Behaviors/Vaccinations
- [Background] Nelson RE, Xie Y, DuVall SL, Butler J, Kamauu AW, Knippenberg K, Schuerch M, Foskett N, LaFleur J. Multiple Sclerosis and Risk of Infection-Related Hospitalization and Death in US Veterans. Int J MS Care. 2015 Sep-Oct;17(5):221-30. doi: 10.7224/1537-2073.2014-035. PMID 26472943
- [Background] Nix EB, Hawdon N, Gravelle S, Biman B, Brigden M, Malik S, McCready W, Ferroni G, Ulanova M. Risk of invasive Haemophilus influenzae type b (Hib) disease in adults with secondary immunodeficiency in the post-Hib vaccine era. Clin Vaccine Immunol. 2012 May;19(5):766-71. doi: 10.1128/CVI.05675-11. Epub 2012 Mar 7. PMID 22398246
- [Background] Olsson T. The new era of multiple sclerosis therapy. J Intern Med. 2014 Apr;275(4):382-6. doi: 10.1111/joim.12196. Epub 2014 Mar 15. No abstract available. PMID 24433367
- [Background] Oreja-Guevara C, Wiendl H, Kieseier BC, Airas L; NeuroNet Study Group. Specific aspects of modern life for people with multiple sclerosis: considerations for the practitioner. Ther Adv Neurol Disord. 2014 Mar;7(2):137-49. doi: 10.1177/1756285613501575. PMID 24587828
- [Background] Orlicka K, Barnes E, Culver EL. Prevention of infection caused by immunosuppressive drugs in gastroenterology. Ther Adv Chronic Dis. 2013 Jul;4(4):167-85. doi: 10.1177/2040622313485275. PMID 23819020
- [Background] Panitch HS. Influence of infection on exacerbations of multiple sclerosis. Ann Neurol. 1994;36 Suppl(Suppl ):S25-8. doi: 10.1002/ana.410360709. PMID 8017885
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Rutschmann OT, McCrory DC, Matchar DB; Immunization Panel of the Multiple Sclerosis Council for Clinical Practice Guidelines. Immunization and MS [RETIRED]: a summary of published evidence and recommendations. Neurology. 2002 Dec 24;59(12):1837-43. doi: 10.1212/wnl.59.12.1837. PMID 12499473
- [Background] Steelman AJ. Infection as an Environmental Trigger of Multiple Sclerosis Disease Exacerbation. Front Immunol. 2015 Oct 19;6:520. doi: 10.3389/fimmu.2015.00520. eCollection 2015. PMID 26539193
- [Background] Vaccines.gov https://www.vaccines.gov/basics/types/index.html
- [Background] Williamson EM, Berger JR. Infection risk in patients on multiple sclerosis therapeutics. CNS Drugs. 2015 Mar;29(3):229-44. doi: 10.1007/s40263-015-0226-2. PMID 25761739
- [Background] Williamson EM, Chahin S, Berger JR. Vaccines in Multiple Sclerosis. Curr Neurol Neurosci Rep. 2016 Apr;16(4):36. doi: 10.1007/s11910-016-0637-6. PMID 26922172
- [Background] Winkelmann A, Loebermann M, Reisinger EC, Hartung HP, Zettl UK. Disease-modifying therapies and infectious risks in multiple sclerosis. Nat Rev Neurol. 2016 Apr;12(4):217-33. doi: 10.1038/nrneurol.2016.21. Epub 2016 Mar 4. PMID 26943779
- [Background] www.cdc.gov Adults with chronic conditions: get vaccinated. Available from https://www.cdc.gov/features/vaccineschronicconditions/index.html. Accessed May 13, 2018.
- [Background] www.ecdc.europa.eu Seasonal influenza vaccines. Influenza vaccination. Available from: http://ecdc.europa.eu/en/healthtopics/seasonal_influenza/vaccines/Pages/ influenza_vaccination.aspx#vaccinationstrategies. Accessed May 13, 2018
- [Background] www.salute.gov Ministero della salute. Vaccinazioni http://www.salute.gov.it/portale/vaccinazioni/homeVaccinazioni.jsp
- [Background] • Yang SH, Hsu C, Cheng AL, Kuo SH (2014) Anti-CD20 monoclonal antibodies and associated viral hepatitis in hematological diseases. World J Hematol, 3(2):29-43